CLINICAL TRIAL: NCT01036490
Title: Structured Exercise in Obese Diabetic Patients With Chronic Kidney Disease
Brief Title: Exercise in Obese Diabetic Patients With Chronic Kidney Disease
Acronym: EX-ODCKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F7264-R
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Results first posted 2016-04-27 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-06

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Control group
- Exercise (Experimental): Exercise Group
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise training for 12 weeks followed by home exercise for 40 weeks
  Arms: Exercise

SUMMARY:
Patients with type 2 diabetes, obesity, and chronic kidney disease are generally physically inactive, have a high mortality rate, and may benefit from an exercise program. This study seeks to determine if a structured exercise program will benefit the heart (improved exercise tolerance, decreased blood pressure) and/or the kidney (decreased protein loss in urine and stabilization of kidney function) and lead to improvements in diabetes, body composition, and quality of life.

DETAILED DESCRIPTION:
Patients with type 2 diabetes, obesity, and chronic kidney disease (CKD) are generally physically inactive, have a high mortality rate, and may benefit from an exercise program. However, there have been no randomized controlled trials to determine the benefits of exercise training in this population. This study seeks to substantiate the hypothesis that increasing energy expenditure by exercise training in the obese diabetic patient with CKD will result in the following benefits:

1. Renal benefits, including reduction in proteinuria and stabilization of glomerular filtration rate (GFR)
2. Cardiovascular benefits, including decreased blood pressure, decreased heart rate, and increased exercise tolerance.
3. Improved glucose control (lower glycated hemoglobin), lipid control (decreased cholesterol with improved atherogenic profile)
4. Improved body composition (weight loss, increased lean body mass and decreased fat mass).
5. Decreased inflammation (assessed by high-sensitivity C-reactive protein), endothelial dysfunction (assessed by flow-mediated dilatation), and oxidative stress (assessed by reduced glutathione).
6. Increased health-related quality of life.

In preparation for this proposal, the investigators performed a 24-week randomized controlled feasibility study comparing aerobic exercise plus optimal medical management to medical management alone in patients with type 2 diabetes, obesity (BMI > 30 kg/m2), and stage 2-4 CKD (eGFR 15-90 mL/min/1.73m2) with persistent proteinuria of > 200 mg/g. Subjects randomized to exercise underwent thrice weekly aerobic training for 6 followed by 18 weeks of supervised home exercise. The primary outcome variable was change in proteinuria. Exercise training resulted in a significant improvement in exercise duration during stress testing which persisted until 24 weeks. This was accompanied by significant decreases in resting systolic blood pressure and 24-hour proteinuria at 24 weeks. No changes were seen in the control group. The investigators concluded that exercise training in obese diabetic patients with CKD is feasible and results in a demonstrable training effect (increased exercise duration and decreased resting blood pressure). Moreover, it may decrease proteinuria and thus have a renoprotective effect.

The investigators now propose a larger-scale randomized controlled trial to determine the effects of exercise on renal functions, cardiovascular fitness, inflammation, and oxidative stress in diabetic patients with CKD. This will be a 52-week randomized study based on the investigators' pilot study design with some modifications. As opposed to the 6-week training period and 18-week home exercise period utilized in the pilot study, subjects randomized to exercise will undergo 12 weeks of intensive exercise training in the exercise laboratory followed by 40 weeks of supervised home exercise training (total duration of study 1 year). Moreover, due to recent recommendations that resistance training be incorporated into exercise training regimens in type 2 diabetic patients, the investigators will incorporate resistance (strength) training in this proposal. The primary outcome variable will be change in proteinuria at 12 and 52 weeks. Secondary outcome variables will be change in albuminuria and estimated glomerular filtration rate (eGFR) at 12 and 52 weeks. In addition, the investigators will measure blood pressure (BP), glycated hemoglobin, lipid profile, C-reactive protein (CRP) levels, body weight and composition, endothelial dysfunction (by flow-mediated dilatation), and Quality of Life (QoL) evaluations. The Index of Coexistent Diseases (ICED) to measure comorbidities to determine if comorbid conditions had any influence on the outcomes of the study. The Center for Epidemiologic Studies Depression Scale (CES-D) will also be used to determine the influence of depression (covariate) on study outcomes and adherence with the study objectives.

This study will directly address the effects of a structured exercise program in a patient population at high risk for cardiovascular complications. The investigators will specifically address the novel idea that exercise will not only improve cardiovascular fitness but will also ameliorate the renal complications resulting from diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus
* CKD Stages 2-4
* BMI > 30
* Persistent proteinuria (urine protein/creatinine > 200 mg/g for > 3 mo)
* On treatment with ACE inhibitor or ARB
* On treatment with aspirin
* On treatment with statin (if LDL > 100)

Exclusion Criteria:

* Symptomatic neuropathy/retinopathy
* Positive stress test due to coronary arterial disease
* Symptomatic cardiovascular disease
* Congestive heart failure (New York Heart Association Class III or IV)
* Chronic obstructive pulmonary disease (FEV1 < 50% predicted and/or requires supplemental oxygen support during exercise)
* Complaints of angina during the stress test
* Cerebrovascular disease/cognitive impairment
* Renal transplant
* Inability to walk on the treadmill
* Any unforeseen illness or disability that would preclude exercise testing or training
* Participation in a formal exercise program within the previous 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-07-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Leehey, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL; Eileen G. Collins, PhD RN, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (1):
- Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Conley MM, McFarlane CM, Johnson DW, Kelly JT, Campbell KL, MacLaughlin HL. Interventions for weight loss in people with chronic kidney disease who are overweight or obese. Cochrane Database Syst Rev. 2021 Mar 30;3(3):CD013119. doi: 10.1002/14651858.CD013119.pub2. PMID 33782940

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the outpatient medical clinics of Hines VA Hospital over the three-year period between January 2011 and January 2014
Groups:
- Exercise: Dietary management plus 12 weeks of combined aerobic and resistance exercise training followed by 40 weeks of supervised home exercise.
- Control: Dietary management alone
Period: Overall Study
Arm/Group | Exercise | Control
Started | 18 | 18
Completed | 14 | 18
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Exercise: 12-week (3 days per week) program of aerobic and resistance training followed by 40 weeks of a home exercise program plus nutritional counseling
- Control: Nutritional counseling alone
- Total: Total of all reporting groups
Arm/Group | Exercise | Control | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (8.7) | 67 (7.5) | 66 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 18 | 18 | 36
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 36.2 (4.8) | 37.4 (4.2) | 37 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Proteinuria
Time Frame: 12 weeks minus baseline
Measure: Median (Inter-Quartile Range); unit: mg/g creatinine
Arm/Group | Exercise | Control
Number analyzed (Participants) | 14 | 18
mg/g creatinine | -34 [-236 to 247] | -133 [-406 to -75]
Statistical Analysis 1: Comparison: Exercise vs Control; Test type: Superiority or Other; p = 0.04, t-test, 2 sided

2. Primary Outcome: Change in Proteinuria
Time Frame: 52 weeks minus baseline
Measure: Median (Inter-Quartile Range); unit: mg/g creatinine
Arm/Group | Exercise | Control
Number analyzed (Participants) | 14 | 18
mg/g creatinine | 15 [-433 to 428] | -66 [-729 to 219]
Statistical Analysis 1: Comparison: Exercise vs Control; Test type: Superiority or Other; p = 0.39, t-test, 2 sided

3. Secondary Outcome: Change in Albuminuria
Time Frame: 12 weeks minus baseline
Measure: Median (Inter-Quartile Range); unit: mg/g creatinine
Arm/Group | Exercise | Control
Number analyzed (Participants) | 14 | 18
mg/g creatinine | -11 [-148 to 203] | -87 [-323 to 1]

4. Secondary Outcome: Change in Albuminuria
Time Frame: 52 weeks minus baseline
Measure: Median (Inter-Quartile Range); unit: mg/g creatinine
Arm/Group | Exercise | Control
Number analyzed (Participants) | 14 | 18
mg/g creatinine | -13 [-372 to 233] | -31 [-598 to 238]

5. Secondary Outcome: Change in Estimated Glomerular Filtration Rate (eGFR)
Time Frame: 12 weeks minus baseline
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Exercise | Control
Number analyzed (Participants) | 14 | 18
mL/min/1.73m^2 | 0.2 (4.7) | -3.4 (8.9)
Statistical Analysis 1: Comparison: Exercise vs Control; Test type: Superiority or Other; p = 0.15, t-test, 2 sided

6. Secondary Outcome: Change in Estimated Glomerular Filtration Rate (eGFR)
Time Frame: 52 weeks minus baseline
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Exercise | Control
Number analyzed (Participants) | 14 | 18
mL/min/1.73m^2 | -2.0 (5.8) | -3.1 (6.0)
Statistical Analysis 1: Comparison: Exercise vs Control; Test type: Superiority or Other; p = 0.58, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Exercise | Control
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

LIMITATIONS AND CAVEATS:
Due to inability to reach our expected target randomization (30 per group), our study may be underpowered to detect differences between the groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No